CLINICAL TRIAL: NCT01691560
Title: A Proof of Concept Study to Evaluate the Efficacy of an Occlusion Based Dentifrice in the Relief of Dentinal Hypersensitivity
Brief Title: Exploratory Study to Evaluate an Occlusion Based Dentifrice in Relief of Dentinal Hypersensitivity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: BioSci Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RH01426
Record Dates: First submitted 2012-09-20; First posted 2012-09-24 (Estimated); Results first posted 2014-05-29 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2013-07

CONDITIONS: Dentine Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 5% calcium sodium phosphosilicate/sodium monofluorophosphate (Experimental): Dentifrice containing 5.0% w/w calcium sodium phosphosilicate with sodium monofluorophosphate containing 1500 parts per million fluoride (ppmF).
  Interventions: Drug: 5% calcium sodium phosphosilicate/ sodium monofluorophosphate dentifrice
- 0% calcium sodium phosphosilicate/sodium monofluorophosphate (Active Comparator): Dentifrice containing 0% w/w calcium sodium phosphosilicate and 1500ppmF as sodium monofluorophosphate
  Interventions: Drug: 0% calcium sodium phosphosilicate/sodium monofluorophosphate dentifrice
- Sodium monofluorophosphate (Active Comparator): Dentifrice containing 1000 ppmF as sodium monofluorophosphate
  Interventions: Drug: Sodium monofluorophosphate dentifrice
- Sodium fluoride (Active Comparator): Dentifrice containing 1100 ppmF as sodium fluoride
  Interventions: Drug: Sodium fluoride dentifrice

INTERVENTIONS:
Drug: 5% calcium sodium phosphosilicate/ sodium monofluorophosphate dentifrice — Dentifrice containing 5.0% w/w calcium sodium phosphosilicate and 1500ppmF as sodium monofluorophosphate
  Arms: 5% calcium sodium phosphosilicate/sodium monofluorophosphate
Drug: 0% calcium sodium phosphosilicate/sodium monofluorophosphate dentifrice — Dentifrice containing 0% w/w calcium sodium phosphosilicate and 1500ppmF as sodium monofluorophosphate
  Arms: 0% calcium sodium phosphosilicate/sodium monofluorophosphate
Drug: Sodium monofluorophosphate dentifrice — Dentifrice containing 1000 ppmF as sodium monofluorophosphate
  Arms: Sodium monofluorophosphate
Drug: Sodium fluoride dentifrice — Dentifrice containing 1100 ppmF as sodium fluoride
  Arms: Sodium fluoride

SUMMARY:
The purpose of this exploratory study is to compare the treatment effect on dentinal hypersensitivity of a tubule occluding dentifrice as measured by Schiff and Tactile sensitivity. This proof of concept study will compare the test dentifrice with three other treatment groups.

DETAILED DESCRIPTION:
This will be a single center, eight week, randomized, controlled, examiner blind, four treatment arm, parallel design, stratified (by maximum baseline Schiff Sensitivity Score of the two selected test teeth), exploratory study in participants with at least two sensitive teeth that meet all the criteria at the Screening and Baseline visit. Participants will be assessed at Baseline, four and eight weeks to monitor clinical efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Participants between 18 and 55 years of age, in good general health, with pre-existing self-reported and clinically diagnosed tooth sensitivity are required for entry into the study
2. Participants will be required to have at least four teeth with facial/cervical erosion, abrasion and/or gingival recession which respond to qualifying evaporative (air) assessment at the Screening visit and have at least two teeth (incisors, canines or pre-molars) demonstrating signs of sensitivity, measured by qualifying tactile threshold (Yeaple ≤ 20 gram (g)) and evaporative (air) (Schiff Sensitivity Score ≥ 2) assessments at the Baseline visit

Exclusion Criteria:

1. Pregnancy: Women who are known to be pregnant or who are intending to become pregnant over the duration of the study.
2. Breast-feeding: Women who are breast-feeding.
3. Medical History: a) Chronic debilitating disease is present b) Chronic disease or other condition is present that is associated with intermittent episodes or constant daily pain, such as arthritis, low back pain, dysmenorrhea, etc.
4. Medications: Daily doses of medication, which in the opinion of the investigator, might interfere with the perception of pain, are being taken. Examples of such medications include analgesics, anticonvulsants, antihistamines that cause marked or moderate sedation, sedatives, tranquilizers, mood-altering and anti-inflammatory drugs.
5. Dentition Exclusions: a) Sensitive teeth not expected to respond to treatment with an over-the- counter dentifrice in the opinion of the investigator. b) Teeth with exposed dentine but with deep, defective or facial restorations, teeth used as abutments for fixed or removable partial dentures, teeth with full crowns, orthodontic bands, extensive caries or cracked enamel. Sensitive teeth with contributing etiologies other than erosion, abrasion or recession of exposed dentine. c) Dental professional hygiene (includes dental prophylaxis, irrigation, and intensive anti-microbial/anti-biotic therapy) within 14 days of the screening visit. d) Presence of dental implants. e) Lip or tongue piercings. f) Periodontal surgical history within the past 6 months or have been scaled /root planed within the past 3 months.
6. Allergy/Intolerance: Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
7. Clinical Study/Experimental Medication: a) Participation in another clinical study or receipt of an investigational drug within 30 days of the screening visit b) Previous participation in this study.
8. Other: Any subject who in the opinion of the investigator, should not participate in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2012-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- BioSci Research America, Las Vegas, Nevada, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site.
Pre-assignment Details: Out of 152 screened participants, 16 did not meet the study criterion while 2 withdrew consent. Hence, a total of 134 participants were randomized into the study.
Groups:
- 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate: Dentifrice containing 5.0% w/w calcium sodium phosphosilicate and 1500 parts per million (ppm) fluoride as sodium monofluorophosphate
- 0% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate: Dentifrice containing 0% w/w calcium sodium phosphosilicate and 1500 ppm fluoride as sodium monofluorophosphate
- Sodium Monofluorophosphate: Dentifrice containing 1000 ppm fluoride as sodium monofluorophosphate
- Sodium Fluoride: Dentifrice containing 1100 ppm fluoride as sodium fluoride
Period: Overall Study
Arm/Group | 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate | 0% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate | Sodium Monofluorophosphate | Sodium Fluoride
Started | 34 | 33 | 34 | 33
Completed | 34 | 33 | 34 | 33
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate: Dentifrice containing 5.0% w/w calcium sodium phosphosilicate and 1500 ppm fluoride as sodium monofluorophosphate
- Total: Total of all reporting groups
Arm/Group | 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate | 0% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate | Sodium Monofluorophosphate | Sodium Fluoride | Total
Number analyzed (Participants) | 34 | 33 | 34 | 33 | 134
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.4 (10.45) | 33.2 (10.13) | 38.2 (8.88) | 36.2 (9.62) | 35.8 (9.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 27 | 22 | 98
  Male | 9 | 9 | 7 | 11 | 36

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Evaporative Air Sensitivity Pain Response on Schiff Sensitivity Scale at Week 4
Description: Response to a constant jet of air applied to hypersensitive teeth was evaluated using a Schiff Sensitivity pain response scale. According to this analog scale, pain response for each individual stimulated tooth ranged from 0 to 3; 0 - participant does not respond to air stimulation, 1 - participant responds to air stimulus but does not request discontinuation of stimulus, 2 - participant responds to air stimulus and request discontinuation of stimulus, 3 - participant responds to air stimulus, considers stimulus to be painful and request discontinuation of stimulus.
Time Frame: Baseline to 4 weeks post administration of study treatment
Population: Intent to Treat (ITT) population: All randomized participants administered with at least one study treatment during the study and provided at least one post baseline assessment of efficacy.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate | Sodium Monofluorophosphate | Sodium Fluoride | 0% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate
Number analyzed (Participants) | 34 | 34 | 33 | 33
Score on a scale | -0.36 [-0.53 to -0.20] | -0.43 [-0.59 to -0.27] | -0.40 [-0.57 to -0.23] | -0.45 [-0.62 to -0.28]
Statistical Analysis 1: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs 0% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.4553, ANCOVA; From ANCOVA model with treatment and baseline included as covariate; Adjusted Mean Difference = 0.09, 95% CI 2-sided [-0.14 to 0.32] — Difference is First named treatment minus Second named treatment that negative difference implies the mean of the second named treatment is larger than that of the first named treatment
Statistical Analysis 2: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs Sodium Monofluorophosphate; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.5689, ANCOVA; From ANCOVA model with treatment and baseline included as covariate; Adjusted mean difference = 0.07, 95% CI 2-sided [-0.16 to 0.30] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs Sodium Fluoride; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.7517, ANCOVA; From ANCOVA model with treatment and baseline included as covariate; Adjusted Mean Difference = 0.04, 95% CI 2-sided [-0.20 to 0.27] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Sodium Monofluorophosphate vs 0% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.8549, ANCOVA; From ANCOVA model with treatment and baseline included as covariate; Adjusted Mean Difference = 0.02, 95% CI 2-sided [-0.21 to 0.25] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Sodium Fluoride vs 0% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.6685, ANCOVA; From ANCOVA model with treatment and baseline included as covariate; Adjusted mean difference = 0.05, 95% CI 2-sided [-0.18 to 0.29] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Sodium Monofluorophosphate vs Sodium Fluoride; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.8031, ANCOVA; Adjusted Mean Difference = -0.03, 95% CI 2-sided [-0.26 to 0.20] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Change From Baseline in Tactile Sensitivity Pain Response (g) at Week 4
Description: Response to increasing force on hypersensitive teeth was evaluated using a Yeaple Probe pain response scale. In tactile sensitivity assessment, an increasing force is applied to hypersensitive tooth until a yes response was recorded or the maximum force was reached.
Time Frame: Baseline to 4 weeks post administration of study treatment
Population: ITT population: All randomized participants administered with at least one study treatment during the study and provided at least one post baseline assessment of efficacy.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate | Sodium Monofluorophosphate | Sodium Fluoride | 0% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate
Number analyzed (Participants) | 34 | 34 | 33 | 33
grams | 7.31 (11.227) | 6.32 (13.045) | 4.09 (4.752) | 3.64 (6.030)
Statistical Analysis 1: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs 0% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.0467, Wilcoxon (Mann-Whitney); Hodges-Lehmann Wilcoxon non-parametric test; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 5] — Difference is First named treatment minus Second named treatment such that a positive difference favors the first named treatment
Statistical Analysis 2: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs Sodium Monofluorophosphate; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.1133, Wilcoxon (Mann-Whitney); Hodges-Lehmann Wilcoxon non-parametric test; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 5] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs Sodium Fluoride; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.2579, Wilcoxon (Mann-Whitney); Hodges-Lehmann Wilcoxon non-parametric test; Median Difference (Final Values) = 0, 95% CI [0 to 5] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Sodium Monofluorophosphate vs 0% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.6149, Wilcoxon (Mann-Whitney); Hodges-Lehmann Wilcoxon non-parametric test; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Sodium Fluoride vs 0% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.3259, Wilcoxon (Mann-Whitney); Hodges-Lehmann Wilcoxon non-parametric test; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 5] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Sodium Monofluorophosphate vs Sodium Fluoride; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.5721, Wilcoxon (Mann-Whitney); Hodges-Lehmann Wilcoxon non-parametric test; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 0] — [estimate comment as in outcome 2, analysis 1]

3. Primary Outcome: Change From Baseline in Evaporative Air Sensitivity Pain Response on Schiff Sensitivity Scale at Week 8
Description: as for outcome 1
Time Frame: Baseline to 8 weeks post administration of study treatment
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate | Sodium Monofluorophosphate | Sodium Fluoride | 0% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate
Number analyzed (Participants) | 34 | 34 | 33 | 33
Score on a scale | -0.55 [-0.78 to -0.33] | -0.43 [-0.66 to -0.20] | -0.43 [-0.66 to -0.20] | -0.92 [-1.15 to -0.68]
Statistical Analysis 1: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs 0% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.0292, ANCOVA; From ANCOVA model with treatment and baseline included as covariate; Adjusted Mean Difference = 0.36, 95% CI 2-sided [0.04 to 0.69] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs Sodium Monofluorophosphate; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.4484, ANCOVA; From ANCOVA model with treatment and baseline included as covariate; Adjusted Mean Difference = -0.12, 95% CI 2-sided [-0.44 to 0.20] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs Sodium Fluoride; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.4537, ANCOVA; From ANCOVA model with treatment and baseline included as covariate; Adjusted Mean Difference = -0.12, 95% CI 2-sided [-0.45 to 0.20] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Sodium Monofluorophosphate vs 0% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.0037, ANCOVA; From ANCOVA model with treatment and baseline included as covariate; Adjusted Mean Difference = 0.49, 95% CI 2-sided [0.16 to 0.81] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Sodium Fluoride vs 0% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.0040, ANCOVA; From ANCOVA model with treatment and baseline included as covariate; Adjusted Mean Difference = 0.48, 95% CI 2-sided [0.16 to 0.81] — Treatment as fixed factor, baseline Schiff score as covariate. Difference is First named treatment minus Second named treatment that negative difference implies the mean of the second named treatment is larger than that of the first named treatment
Statistical Analysis 6: Comparison: Sodium Monofluorophosphate vs Sodium Fluoride; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.9974, ANCOVA; From ANCOVA model with treatment and baseline included as covariate; Adjusted Mean Difference = 0.00, 95% CI 2-sided [-0.32 to 0.32] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Change From Baseline in Tactile Sensitivity Pain Response (g) at Week 8
Description: as for outcome 2
Time Frame: Baseline to 8 weeks post administration of study treatment
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate | Sodium Monofluorophosphate | Sodium Fluoride | 0% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate
Number analyzed (Participants) | 34 | 34 | 33 | 33
grams | 10.15 (15.100) | 5.88 (11.512) | 4.39 (5.556) | 11.97 (16.486)
Statistical Analysis 1: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs 0% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.8861, Wilcoxon (Mann-Whitney); Hodges-Lehmann Wilcoxon non-parametric test; Median Difference (Final Values) = 0, 95% CI 2-sided [-5 to 5] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs Sodium Monofluorophosphate; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.0641, Wilcoxon (Mann-Whitney); Hodges-Lehmann Wilcoxon non-parametric test; Median Difference (Final Values) = 0, 95% CI 2-sided [0 to 5] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs Sodium Fluoride; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.1831, Wilcoxon (Mann-Whitney); Hodges-Lehmann Wilcoxon non-parametric test; Median Difference (Final Values) = 0, 95% CI [0 to 5] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Sodium Monofluorophosphate vs 0% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.0871, Wilcoxon (Mann-Whitney); Hodges-Lehmann Wilcoxon non-parametric test; Median Difference (Final Values) = 0, 95% CI 2-sided [-10 to 0] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Sodium Fluoride vs 0% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.1690, Wilcoxon (Mann-Whitney); Hodges-Lehmann Wilcoxon non-parametric test; Median Difference (Final Values) = 0, 95% CI 2-sided [-10 to 0] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Sodium Monofluorophosphate vs Sodium Fluoride; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.3829, Wilcoxon (Mann-Whitney); Hodges-Lehmann Wilcoxon non-parametric test; Median Difference (Final Values) = 0, 95% CI 2-sided [-5 to 0] — [estimate comment as in outcome 2, analysis 1]

5. Primary Outcome: Change From Baseline in Evaporative Air Sensitivity Response on a Visual Rating Scale (VRS) at Week 4
Description: Participants rated the intensity of their response to the stimulus using a 10 point Visual rating scale of 1 (no Pain) to 10 (intense pain).
Time Frame: Baseline to 4 weeks post administration of study treatment
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate | Sodium Monofluorophosphate | Sodium Fluoride | 0% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate
Number analyzed (Participants) | 34 | 34 | 33 | 33
Score on a scale | -1.22 [-1.76 to -0.69] | -1.07 [-1.60 to -0.55] | -1.35 [-1.89 to -0.81] | -1.25 [-1.80 to -0.71]
Statistical Analysis 1: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs 0% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.9421, ANCOVA; ANCOVA with treatment and Schiff stratification as factors and baseline VRS as covariate; Adjusted Mean Difference = 0.03, 95% CI 2-sided [-0.74 to 0.80] — Difference is first named treatment minus second named treatment that a negative difference implies the mean of second named treatment is larger than that of the first named treatment
Statistical Analysis 2: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs Sodium Monofluorophosphate; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.6918, ANCOVA; ANCOVA with treatment and Schiff stratification as factors and baseline VRS as covariate; Adjusted Mean Difference = -0.15, 95% CI 2-sided [-0.90 to 0.60] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs Sodium Fluoride; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.7421, ANCOVA; From ANCOVA with treatment and Schiff stratification as factors and baseline VRS as covariate; Adjusted Mean Difference = 0.13, 95% CI 2-sided [-0.63 to 0.88] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Sodium Monofluorophosphate vs 0% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.6433, ANCOVA; From ANCOVA with treatment and Schiff stratification as factors and baseline VRS as covariate; Adjusted Mean Difference = 0.18, 95% CI 2-sided [-0.58 to 0.94] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: Sodium Fluoride vs 0% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.8010, ANCOVA; From ANCOVA with treatment and Schiff stratification as factors and baseline VRS as covariate; Adjusted Mean Difference = -0.10, 95% CI 2-sided [-0.86 to 0.67] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 6: Comparison: Sodium Monofluorophosphate vs Sodium Fluoride; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.4692, ANCOVA; From ANCOVA with treatment and Schiff stratification as factors and baseline VRS as covariate; Adjusted Mean Difference = 0.28, 95% CI 2-sided [-0.48 to 1.03] — [estimate comment as in outcome 5, analysis 1]

6. Primary Outcome: Change From Baseline in Evaporative Air Sensitivity Response on VRS at Week 8
Description: Participants rated the intensity of their response to the stimulus using a 10 point VRS of 1 (no Pain) to 10 (intense pain).
Time Frame: Baseline to 8 weeks post administration of study treatment
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate | Sodium Monofluorophosphate | Sodium Fluoride | 0% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate
Number analyzed (Participants) | 34 | 34 | 33 | 33
Score on a scale | -1.76 [-2.35 to -1.17] | -1.22 [-1.81 to -0.63] | -1.31 [-1.90 to -0.71] | -2.06 [-2.67 to -1.46]
Statistical Analysis 1: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs 0% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.4797, ANCOVA; From ANCOVA with treatment and Schiff stratification as factors and baseline VRS as covariate; Adjusted Mean Difference = 0.31, 95% CI 2-sided [-0.55 to 1.16] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 2: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs Sodium Monofluorophosphate; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.2023, ANCOVA; From ANCOVA with treatment and Schiff stratification as factors and baseline VRS as covariate; Adjusted Mean Difference = -0.54, 95% CI 2-sided [-1.37 to 0.29] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 3: Comparison: 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate vs Sodium Fluoride; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.2917, ANCOVA; From ANCOVA with treatment and Schiff stratification as factors and baseline VRS as covariate; Adjusted Mean Difference = -0.45, 95% CI 2-sided [-1.29 to 0.39] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 4: Comparison: Sodium Monofluorophosphate vs 0% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.0503, ANCOVA; From ANCOVA with treatment and Schiff stratification as factors and baseline VRS as covariate; Adjusted Mean Difference = 0.85, 95% CI 2-sided [0.00 to 1.69] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 5: Comparison: Sodium Fluoride vs 0% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.0811, ANCOVA; From ANCOVA with treatment and Schiff stratification as factors and baseline VRS as covariate; Adjusted Mean Difference = 0.76, 95% CI 2-sided [-0.09 to 1.61] — [estimate comment as in outcome 5, analysis 1]
Statistical Analysis 6: Comparison: Sodium Monofluorophosphate vs Sodium Fluoride; Null hypothesis considered change from baseline to be same for treatments in comparison; Test type: Superiority or Other; p = 0.8322, ANCOVA; From ANCOVA with treatment and Schiff stratification as factors and baseline VRS as covariate; Adjusted Mean Difference = 0.09, 95% CI 2-sided [-0.75 to 0.93] — [estimate comment as in outcome 5, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were collected collected from the start of the investigational product (or washout product), and until 5 days following last administration of the investigational product.
Arm/Group | 5% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate | 0% Calcium Sodium Phosphosilicate/ Sodium Monofluorophosphate | Sodium Monofluorophosphate | Sodium Fluoride
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/33 | 0/34 | 0/33
Other Adverse Events (participants affected / at risk) | 0/34 | 0/33 | 0/34 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.